CLINICAL TRIAL: NCT03439488
Title: A Multipart Phase 1, Double-Blind, Randomized, Placebo-Controlled, First-in-Human, Study of Orally Administered JNJ-440 to Evaluate the Safety, Tolerability, and Pharmacokinetics After Single Ascending Doses Including Food Effect Evaluation (Part 1); After Multi-Day Dosing (Part 2) in Healthy Subjects; and After Multiple (Ascending) Doses in Subjects With Chronic Hepatitis B (Part 3)
Brief Title: A Study of Orally Administered JNJ-440 to Evaluate the Safety, Tolerability, and Pharmacokinetics After Single Ascending Doses Including Food Effect Evaluation; After Multi-Day Dosing in Healthy Participants; and After Multiple (Ascending) Doses in Participants With Chronic Hepatitis B
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Alios Biopharma Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Other
Other Study IDs: JNJ-440-1301; JNJ-440-1301 (Other: Alios Biopharma Inc.); 2017-004657-17 (EudraCT Number)
Record Dates: First submitted 2018-01-23; First posted 2018-02-20 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Chronic Hepatitis B
Keywords: First in Human; Healthy Volunteers; Hepatitis B Virus; JNJ-64530440
MeSH Terms: conditions — Hepatitis B, Chronic; Hepatitis B

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Part 1 (Healthy Participants): Single Ascending Dose (SAD) (Experimental): Participants in Cohorts 1 to 5 and 3 optional cohorts (Cohorts 6, 7 and 10) will receive a single dose of JNJ-440/placebo on Day 1. Two cohorts will receive a second dose of JNJ-440/placebo in a fed state (participants from Cohort 3 will also participate in Cohort 8) or as an alternative JNJ-440 formulation (participants from Cohort 2 will also participate in optional Cohort 9) after a washout window of at least 10 days. In Cohorts 1 to 4, study drug will be administered under fasted conditions; in the remaining cohorts, study drug will be administered under fasted/fed conditions depending on the results of the food effect evaluation.
  Interventions: Drug: JNJ-440; Drug: Placebo
- Part 2 (Healthy Participants): Multiple Ascending Dose (MAD) (Experimental): Participants in Cohorts 1 and 2 will receive a once daily dose of JNJ-440/placebo for the duration of 7 days under fasted or fed conditions. Participants in an optional cohort (Cohort 3) may receive a once daily or twice daily dose of JNJ-440/placebo for the duration of 7 or 14 days under fasted or fed conditions. The starting dose for Cohort 1 in Part 2 will be determined by the Sponsor in consultation with the Principal Investigator based on the data from Part 1. Dose escalation will be performed only after review of safety and pharmacokinetic (PK) data after a minimum of 7 days of study drug administration.
  Interventions: Drug: JNJ-440; Drug: Placebo
- Part 3 (Chronic Hepatitis B [CHB] Participants): MAD (Experimental): Participants in Cohorts 1 and 2 and 3 optional cohorts (Cohorts 3, 4, and 5) will receive multiple ascending doses of JNJ-440/placebo once daily or twice daily for 28 days under fed or fasted conditions. The starting dose and formulation for Cohort 1 will be determined based on the review of available data in healthy participants from Part 1 (SAD) and Part 2 (MAD). Dose escalation will be performed only after review of safety, tolerability, and PK data after a minimum of 14 days of study drug administration from at least 8 CHB participants.
  Interventions: Drug: JNJ-440; Drug: Placebo

INTERVENTIONS:
Drug: JNJ-440 — JNJ-440 will be administered as oral tablets in Parts 1, 2 and 3. JNJ-440 may be provided as oral solution in a cohort in Part 1.
  Other Names: JNJ-64530440 or ALS-003440
Drug: Placebo — Matching placebo as oral tablets will be administered in Parts 1, 2 and 3.

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of JNJ-440 in healthy and Chronic Hepatitis B (CHB) participants after single and multiple doses; and to evaluate the pharmacokinetic (PK) of JNJ-440 in healthy participants and in CHB participants following single and multiple dose regimens, administered alone (healthy participants and CHB participants).

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria for Healthy Participants:

* Female participants (except for postmenopausal women) must have a negative pregnancy test at screening and on Day -1
* Participants must have a body mass index (BMI; weight in kilogram [kg] divided by the square of height in meters) of 18.0 to 30.0 kilogram per meter square (kg/m^2), extremes included
* Participants must agree not to donate blood during the study and for at least 1 month after the completion of study drug administration

Inclusion Criteria for Participants with Chronic Hepatitis B (CHB):

* Participant must have CHB infection documented by: (a) Serum hepatitis B surface antigen (HBsAg) positive at screening and at least 6 months prior to screening; (b) Serum antibody immunoglobulin M (IgM) anti-HBc antibody negative at screening
* Participants must currently not be receiving any CHB treatment at screening, that is, have never received treatment with hepatitis B virus (HBV) antiviral medicines, nucleos(t)ide analog (NAs), interferon (IFN) products, or investigational anti-HBV agents, OR Have not been on treatment with HBV antiviral medicines, NAs, or IFN products within 6 months prior to baseline (first intake of study drugs)

Exclusion Criteria:

Exclusion Criteria for Healthy Participants:

* Participants with a past history of cardiac arrhythmias (example, extrasystoli, tachycardia at rest), history of risk factors for Torsade de Pointes syndrome (example, hypokalemia, family history of long QT Syndrome) or history or other clinical evidence of significant or unstable cardiac disease (example, angina, congestive heart failure, myocardial infarction, diastolic dysfunction, significant arrhythmia, coronary heart disease, and/or clinically significant electrocardiogram [ECG] abnormalities), moderate to severe valvular disease or uncontrolled hypertension at screening. Any evidence of heart block or bundle branch block is also exclusionary
* Participants with any history of confirmed clinically significant skin disease such as, but not limited to, dermatitis, eczema, drug rash, psoriasis, food allergy, and urticarial
* Participants with a history of confirmed clinically significant drug allergy such as, but not limited to, sulfonamides and penicillins, or drug allergy witnessed in previous studies with experimental drugs

Exclusion Criteria for Participants with CHB:

* Participant with positivity of anti-HBs antibodies
* Participants with current hepatitis D virus (HDV) infection (confirmed by HDV antibody) at screening

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 130 (Actual)
Dates: Start 2018-03-26 (Actual); Primary Completion 2019-10-10 (Actual); Study Completion 2019-10-10 (Actual)

PRIMARY OUTCOMES:
Parts 1, 2, and 3: Number of Participants With Adverse Events (AEs) as a Measure of Safety and Tolerability | Approximately up to 8 weeks
  Number of participants with AE (any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship) will be reported.
Parts 1, 2, and 3: Number of Participants With Clinically Significant Changes in Physical Examination (Body Weight Measurement and Skin Examination) | Approximately up to 8 weeks
  A symptom directed physical examination (including body weight measurement and skin examination) will be performed to further assess number of participants with clinically significant changes.
Parts 1, 2, and 3: Number of Participants With Clinically Significant Changes in Vital Signs | Approximately up to 8 weeks
  Number of participants with clinically significant changes in the vital signs will be reported.
Parts 1, 2, and 3: Number of Participants With ECG Abnormalities | Approximately up to 8 weeks
  Number of participants with electrocardiogram (ECG) abnormalities will be reported.
Parts 1, 2, and 3: Number of Participants With Holter Monitoring Abnormalities | Up to 24 hours post-dose on Day 1
  Number of participants with Holter monitoring abnormalities will be reported.
Parts 1, 2, and 3: Number of Participants With Clinical Laboratory Abnormalities | Approximately up to 8 weeks
  Number of participants with clinical laboratory abnormalities will be reported.
Part 1: Maximum Observed Plasma Concentration (Cmax) | Day 1 (predose and at 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 18, 24, 36, 48, 72, 96, and 120 hours postdose)
  The Cmax is the maximum observed plasma concentration.
Part 1: Area Under the Plasma Concentration-Time Curve From Time Zero to Last Quantifiable Time (AUC [0-last]) | Day 1 (predose and at 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 18, 24, 36, 48, 72, 96, and 120 hours postdose)
  The AUC (0-last) is the area under the plasma concentration-time curve from time zero to last quantifiable time.
Part 1: Area Under the Plasma Concentration-Time Curve From Time Zero to Infinite Time (AUC[0-infinity]) | Day 1 (predose and at 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 18, 24, 36, 48, 72, 96, and 120 hours postdose)
  The AUC (0-infinity) is the area under the plasma concentration-time curve from time zero to infinite time, calculated as the sum of AUC(last) and C(last)/lambda(z); wherein AUC(last) is area under the plasma concentration-time curve from time zero to last quantifiable time, C(last) is the last observed quantifiable concentration, and lambda(z) is elimination rate constant.
Part 3: Maximum Observed Plasma Concentration (Cmax) | Day 1 (predose, and at 0.5, 1, 2, 4, 8, and 12 hours post dose), morning predose on Days 2, 15 and 21, and Day 28 (predose, and at 0.5, 1, 2, 4, 8, and 12 hours postdose; 24 hours postdose [once daily {QD} dosing only])
  The Cmax is the maximum observed plasma concentration.
Part 3: Observed Plasma Concentration From Time 0 to tau Hours Postdose (C[0-tau]) | Day 1 (predose, and at 0.5, 1, 2, 4, 8, and 12 hours post dose), morning predose on Days 2, 15 and 21, and Day 28 (predose, and at 0.5, 1, 2, 4, 8, and 12 hours postdose; 24 hours postdose [QD dosing only])
  C(0-tau) is defined as the observed plasma concentration from time 0 to tau hours postdose (tau = dosing interval).
Part 3: Area Under the Curve From Time Zero to End of Dosing Interval (AUC[0-tau]) | Day 1 (predose, and at 0.5, 1, 2, 4, 8, and 12 hours post dose), morning predose on Days 2, 15 and 21, and Day 28 (predose, and at 0.5, 1, 2, 4, 8, and 12 hours postdose; 24 hours postdose [QD dosing only])
  The AUCtau is the measure of the plasma drug concentration from time zero to end of dosing interval. It is used to characterize drug absorption.

SECONDARY OUTCOMES:
Part 1: Ratio of Cmax Values Between Test and Reference Ratio (Cmax, test/reference) for Different Dosage Forms | Day 1 (predose and at 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 18, 24, 36, 48, 72, 96, and 120 hours postdose)
  Ratio Cmax, test/reference is the ratio of individual Cmax values between test and reference treatment. Test = JNJ-440 in oral solution (Cohort 9) or tablet (Cohort 10), and reference = JNJ-440 in fasted conditions (Cohort 2 or Cohort 4-7 [depending on dose], respectively).
Part 1: Ratio of AUC(0-last) Values Between Test and Reference (Ratio AUC[0-last],test/reference) for Different Dosage Forms | Day 1 (predose and at 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 18, 24, 36, 48, 72, 96, and 120 hours postdose)
  Ratio AUC(0-last),test/ref is the ratio of individual AUC(0-last) values between test and reference treatment. Test = JNJ-440 in oral solution (Cohort 9) or tablet (Cohort 10), and reference = JNJ-440 in fasted conditions (Cohort 2 or Cohort 4-7 [depending on dose], respectively).
Part 1: Ratio of AUC(0-infinity) Values Between Test and Reference (Ratio AUC[0-infinity], test/reference) for Different Dosage Forms | Day 1 (predose and at 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 18, 24, 36, 48, 72, 96, and 120 hours postdose)
  Ratio AUC(0-infinity),test/ref is the ratio of individual AUC(0-infinity) values between test and reference treatment. Test = JNJ-440 in oral solution (Cohort 9) or tablet (Cohort 10), and ref = JNJ-440 in fasted conditions (Cohort 2 or Cohort 4-7 [depending on dose], respectively).
Part 1: Ratio of Cmax Values Between Fed and Fasted (Ratio Cmax, test/reference) Conditions | Day 1 (predose and at 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 18, 24, 36, 48, 72, 96, and 120 hours postdose)
  Ratio Cmax, test/reference is the ratio of individual Cmax values between test and reference treatment. Test = JNJ-440 in fed conditions (Cohort 8), and reference = JNJ-440 in fasted conditions (Cohort 3).
Part 1: Ratio of AUC(0-last) Values Between Fed and Fasted (Ratio AUC[0- last],test/reference) | Day 1 (predose and at 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 18, 24, 36, 48, 72, 96, and 120 hours postdose)
  Ratio AUC(0-last),test/ref is the ratio of individual AUC(0-last) values between test and reference treatment. Test = JNJ-440 in fed conditions (Cohort 8), and ref = JNJ-440 in fasted conditions (Cohort 3).
Part 1: Ratio of AUC(0-infinity) Values Between Fed and Fasted (Ratio AUC[0-infinity], test/reference) | Day 1 (predose and at 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 18, 24, 36, 48, 72, 96, and 120 hours postdose)
  Ratio AUC(0-infinity),test/ref is the ratio of individual AUC(0- infinity) values between test and reference treatment. Test = JNJ-440 in fed conditions (Cohort 8), and ref = JNJ-440 in fasted conditions (Cohort 3).
Part 3: Mean Change from Baseline in HBV DNA Levels | Baseline up to Day 56
  Changes of hepatitis B virus (HBV) deoxyribonucleic acid (DNA) levels as assessed by mean change from baseline in HBV DNA will be evaluated.
Part 3: Percentage of Participants with HBV DNA Levels and Undetectable HBV DNA | Baseline up to Day 56
  Percentage of participants with HBV DNA levels such as less than (<) 100 international units per milliliter (IU/mL) and undetectable HBV DNA will be evaluated.
Part 3: Change From Baseline in Hepatitis B Surface Antigen (HBsAg) Levels | Baseline up to Day 56
  The difference of HBsAg levels from baseline will be evaluated.
Part 3: Change From Baseline in Hepatitis B e Antigen (HBeAg) Levels | Baseline up to Day 56
  The difference of HBeAg levels from baseline will be evaluated.
Part 3: Relationship Between Plasma Concentration and Antiviral Activity | Up to Day 56
  The potential association between antiviral activity (like HBV DNA or HBsAg or HBeAg) and plasma concentration of JNJ-440 will be assessed.
Part 3: Relationship Between Plasma Concentration and Select AEs or Laboratory Changes | Up to Day 56
  The potential association between select AEs or laboratory changes and plasma concentration of JNJ-440 may be assessed. Based on the clinically relevant AEs or laboratory changes during the study, this analysis may be performed.
Part 3: Change From Baseline in HBV DNA (Antiviral Activity) in Chronic Hepatitis B (CHB) Participants with Sequence Variations in the HBV Genome | Baseline up to Day 56
  Sequence variations in the HBV genome will be assessed by sequencing of the viral genome. Antiviral activity will be assessed by measuring change from baseline in HBV DNA concentration and compared between participants with and without HBV sequence variations.
Part 3: Number of Participants with Emergence of Treatment Associated Mutations in the HBV Genome | Baseline up to Day 29
  Treatment induced emerging mutations will be assessed by comparing the HBV genome sequence obtained at baseline with sequences obtained post-baseline.
Parts 1, 2, and 3: Relationship Between JNJ-440 Plasma Concentrations and Time-Matched Change from Baseline QTcF | Approximately up to 18 weeks
  The relationship between plasma levels of JNJ-440 and Q-T interval corrected for heart rate according to Fridericia's formula (QTcF) exposure response relationship will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Jeysen Yogaratnam, Study Director — Alios Biopharma Inc.
Locations (7):
- Republican Clinical Hospital, Chisnau, Moldova
- Auckland Clinical Services, Auckland, New Zealand
- South Korea (2):
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
- Thailand (2):
  - Research Unit of Hepatitis and Liver Cancer, Department.Biochemistry, Faculty of Medicine King Chulalongkorn Memorial Hospital, Bangkok
  - Srinagarind Hospital Department of Gastroenterology, Faculty of Medicine, Khon Kaen University, Khon Kaen
- Limited Liability Company "ARENSIA EXPLORATORY MEDICINE", Kapitanavka, Ukraine

REFERENCES:
- [Derived] Kakuda TN, Yogaratnam JZ, Westland C, Gane EJ, Schwabe C, Vuong J, Patel M, Snoeys J, Talloen W, Lenz O, Fry J, Chanda S, van Remoortere P. Pharmacokinetics, safety and tolerability of single- and multiple-ascending doses of JNJ-64530440, a novel hepatitis B virus capsid assembly modulator, in healthy volunteers. Antivir Ther. 2021 Jan-Feb;26(1-2):13-24. doi: 10.1177/13596535211044331. Epub 2021 Sep 23. PMID 35485346
- [Derived] Gane EJ, Schwabe C, Berliba E, Tangkijvanich P, Jucov A, Ghicavii N, Verbinnen T, Lenz O, Talloen W, Kakuda TN, Westland C, Patel M, Yogaratnam JZ, Dragone L, Van Remoortere P. Safety, antiviral activity and pharmacokinetics of JNJ-64530440, a novel capsid assembly modulator, as 4 week monotherapy in treatment-naive patients with chronic hepatitis B virus infection. J Antimicrob Chemother. 2022 Mar 31;77(4):1102-1110. doi: 10.1093/jac/dkab491. PMID 35040959